CLINICAL TRIAL: NCT05898139
Title: Describe to Better Understand, the Mealtime of People With Parkinson's Disease Dependent on Food Intake
Acronym: AideAlimPark
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0527; 2023-A00393-42 (Other: ID-RCB)
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Deglutition Disorders
Keywords: Dysphagia; Assistance feeding; Parkinson disease; Caregivers; Mealtime
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assisting (caregiver) / aided (patient with Parkinsonian syndrome) dyad: The dyad will be filmed during a meal and an interview with the sick person and his caregiver will be carried out independently. Between 15 days and a month after the first visit, excerpts from the film will be presented and commented by the dyad according to the technique of self-confrontation

SUMMARY:
The main objective is to describe strategies (verbal, non-verbal (gesture, intonation), and environmental), designed and used by the assisting/aided dyad to feed a dysphagic dependent person by articulating the safe and hedonic dimensions in the context of Parkinson's disease or atypical parkinsonian syndrome during a meal

DETAILED DESCRIPTION:
It is described in the literature that being helped for the meal disrupts the pre-oral phase in the visual and proprioceptive afferences received by the sick person to prepare neurologically the other phases of swallowing. In cases of dysphagia, regardless of the cause, the need for food assistance is correlated with higher mortality and an increased risk of pneumonia. Thus, whether at home or in an establishment, human help is often put in place to facilitate the time of the meal, make it more effective (limitation of the duration of the meal, maximization of the nutritional amounts ingested) and safe (prevention of the occurrence of wrong driving). Our hypothesis is that representations about food and aid at meal times, as well as the attitudes of both the helper and the helped, are factors influencing the realization of an adapted human aid when eating a meal in a dependent person. An observation of a meal during a hospitalization and an interview with the sick person and his caregiver are carried out independently. Between 15 days and a month after the first visit, excerpts from the film will be presented and commented by the dyad according to the technique of self-confrontation. A report of the thematic elements identified during the interviews will be proposed for validation by the dyad. This visit can be made during a scheduled appointment in the hospital, by videoconference or at home if the participants do not have access to a videoconference system.

ELIGIBILITY:
For patients:

Inclusion Criteria:

* Patient with typical or atypical Parkinsonian syndrome, collected in the medical record
* Indication of swallowing disorders or dysphagia, according to item 2.3 chewing and swallowing, part II of the MSD/UPDRS scale or collection in the medical record
* Person dependent on food (according to MDS/UPDRS - food tasks item, part II, 2.4 ≥ 2, to be help to cut food punctually
* Having a usual caregiver present for the meal.
* Affiliated person or beneficiary of a social security scheme.
* Free, informed, written and signed consent by participant and investigator (no later than the day of inclusion and prior to any review required by the research)

Exclusion Criteria:

* Individuals whose cognitive state does not allow simple questions to be answered, as judged by the neurologist
* Person fed exclusively by enteral nutrition.
* Patient who refuses to be filmed

For caregivers:

Inclusion Criteria:

* caregiver of the patient for at least 2 months for the taking of meal
* Person with French language to answer the questions of the interview

Exclusion Criteria:

* Patient who refuses to be filmed
* Protected patient: under guardianship, trusteeship or other legal protection, deprived of freedom by judicial or administrative decision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with typical or atypical parkinsonian syndrome and their caregiver
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Strategies description | 13 months
  Description of the strategies designed and used by the assisting/aided dyad to feed dysphagic patients to perform the hand-to-mouth gesture in the context of Parkinson's disease or atypical parkinsonian syndrome during a meal, using filmed data and semi-directional interviews.

SECONDARY OUTCOMES:
Description of the perception of meal time, patient's point of view | 13 months
  Thematic analysis of the perception of meal timing, diet, meal assistance for the sick person.
Description of the perception of meal time, helper's point of view | 13 months
  Thematic analysis of the perception of meal timing, diet, meal assistance for the caregiver
Description of quality of life related to meal time | 13 months
  Identify factors that contribute to and detract from meal-related quality of life satisfaction.
Identification of specific needs for educational programmes | 13 months
  Identify the needs of carers to adapt or place specific educational programmes
Description of strategies put in place during meal time | 13 months
  Overview of the strategies put in place to promote a compromise between nutritional, safety and hedonic objectives

CONTACTS AND LOCATIONS:
Overall Officials: Margherita FABBRI, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Parkinson center, Toulouse, Haute-Garonne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batchelor-Murphy MK, McConnell ES, Amella EJ, Anderson RA, Bales CW, Silva S, Barnes A, Beck C, Colon-Emeric CS. Experimental Comparison of Efficacy for Three Handfeeding Techniques in Dementia. J Am Geriatr Soc. 2017 Apr;65(4):e89-e94. doi: 10.1111/jgs.14728. Epub 2017 Feb 6. PMID 28165618
- [Background] Cosentino G, Avenali M, Schindler A, Pizzorni N, Montomoli C, Abbruzzese G, Antonini A, Barbiera F, Benazzo M, Benarroch EE, Bertino G, Cereda E, Clave P, Cortelli P, Eleopra R, Ferrari C, Hamdy S, Huckabee ML, Lopiano L, Marchese Ragona R, Masiero S, Michou E, Occhini A, Pacchetti C, Pfeiffer RF, Restivo DA, Rondanelli M, Ruoppolo G, Sandrini G, Schapira AHV, Stocchi F, Tolosa E, Valentino F, Zamboni M, Zangaglia R, Zappia M, Tassorelli C, Alfonsi E. A multinational consensus on dysphagia in Parkinson's disease: screening, diagnosis and prognostic value. J Neurol. 2022 Mar;269(3):1335-1352. doi: 10.1007/s00415-021-10739-8. Epub 2021 Aug 21. PMID 34417870
- [Background] Fabbri M, Coelho M, Abreu D, Guedes LC, Rosa MM, Godinho C, Cardoso R, Guimaraes I, Antonini A, Zibetti M, Lopiano L, Ferreira JJ. Dysphagia predicts poor outcome in late-stage Parkinson's disease. Parkinsonism Relat Disord. 2019 Jul;64:73-81. doi: 10.1016/j.parkreldis.2019.02.043. Epub 2019 Mar 2. PMID 30902528
- [Background] Flora L, Berkesse A, Payot A, Dumez V, Karazivan P. [THE APPLICATION OF AN INTEGRATED MODEL OF PARTNERSHIP- PATIENT IN THE PROFESSIONALS OF THE HEALTH TRAINING: TOWARDS NEW ONE HUMANIST PARADIGM AND ETHICS OF CO-CONSTRUCTION KNOWLEDGES IN HEALTH]. J Int Bioethique Ethique Sci. 2016 Mar-Jun;27(1-2):59-72, 228. French. PMID 27305793
- [Background] Howells SR, Cornwell PL, Ward EC, Kuipers P. Living with Dysphagia in the Community: Caregivers "do whatever it takes.". Dysphagia. 2021 Feb;36(1):108-119. doi: 10.1007/s00455-020-10117-y. Epub 2020 Apr 24. PMID 32333212
- [Background] Leow LP, Huckabee ML, Anderson T, Beckert L. The impact of dysphagia on quality of life in ageing and Parkinson's disease as measured by the swallowing quality of life (SWAL-QOL) questionnaire. Dysphagia. 2010 Sep;25(3):216-20. doi: 10.1007/s00455-009-9245-9. Epub 2009 Aug 13. PMID 19680723
- [Background] Liu W, Williams K, Batchelor-Murphy M, Perkhounkova Y, Hein M. Eating performance in relation to intake of solid and liquid food in nursing home residents with dementia: A secondary behavioral analysis of mealtime videos. Int J Nurs Stud. 2019 Aug;96:18-26. doi: 10.1016/j.ijnurstu.2018.12.010. Epub 2019 Jan 3. PMID 30660444
- [Background] Liu W, Batchelor M, Williams K. Ease of use, feasibility and inter-rater reliability of the refined Cue Utilization and Engagement in Dementia (CUED) mealtime video-coding scheme. J Adv Nurs. 2020 Dec;76(12):3609-3622. doi: 10.1111/jan.14548. Epub 2020 Sep 30. PMID 32996629
- [Background] Liu W, Tripp-Reimer T, Williams K, Shaw C. Facilitators and barriers to optimizing eating performance among cognitively impaired older adults: A qualitative study of nursing assistants' perspectives. Dementia (London). 2020 Aug;19(6):2090-2113. doi: 10.1177/1471301218815053. Epub 2018 Nov 27. PMID 30482090
- [Background] Miller N, Noble E, Jones D, Burn D. Hard to swallow: dysphagia in Parkinson's disease. Age Ageing. 2006 Nov;35(6):614-8. doi: 10.1093/ageing/afl105. PMID 17047007
- [Background] Perry SE, Borders JC, Dakin AE, Troche MS. Characterizing Quality of Life in Caregivers of People with Parkinson's Disease and Dysphagia. Dysphagia. 2022 Jun;37(3):523-532. doi: 10.1007/s00455-021-10299-z. Epub 2021 May 15. PMID 33991229
- [Background] Pflug C, Bihler M, Emich K, Niessen A, Nienstedt JC, Flugel T, Koseki JC, Plaetke R, Hidding U, Gerloff C, Buhmann C. Critical Dysphagia is Common in Parkinson Disease and Occurs Even in Early Stages: A Prospective Cohort Study. Dysphagia. 2018 Feb;33(1):41-50. doi: 10.1007/s00455-017-9831-1. Epub 2017 Aug 21. PMID 28828545
- [Background] Pomey MP, Flora L, Karazivan P, Dumez V, Lebel P, Vanier MC, Debarges B, Clavel N, Jouet E. [The Montreal model: the challenges of a partnership relationship between patients and healthcare professionals]. Sante Publique. 2015 Jan-Feb;27(1 Suppl):S41-50. French. PMID 26168616
- [Background] Pu D, Yiu EML, Chan KMK. Factors associated with signs of aspiration in older adults: A prospective study. Geriatr Nurs. 2020 Sep-Oct;41(5):635-640. doi: 10.1016/j.gerinurse.2020.03.019. Epub 2020 May 10. PMID 32402573
- [Background] Schindler A, Pizzorni N, Cereda E, Cosentino G, Avenali M, Montomoli C, Abbruzzese G, Antonini A, Barbiera F, Benazzo M, Benarroch E, Bertino G, Clave P, Cortelli P, Eleopra R, Ferrari C, Hamdy S, Huckabee ML, Lopiano L, Marchese-Ragona R, Masiero S, Michou E, Occhini A, Pacchetti C, Pfeiffer RF, Restivo DA, Rondanelli M, Ruoppolo G, Sandrini G, Schapira A, Stocchi F, Tolosa E, Valentino F, Zamboni M, Zangaglia R, Zappia M, Tassorelli C, Alfonsi E. Consensus on the treatment of dysphagia in Parkinson's disease. J Neurol Sci. 2021 Nov 15;430:120008. doi: 10.1016/j.jns.2021.120008. Epub 2021 Sep 27. PMID 34624796
- [Background] Shune SE, Namasivayam-MacDonald AM. Swallowing Impairments Increase Emotional Burden in Spousal Caregivers of Older Adults. J Appl Gerontol. 2020 Feb;39(2):172-180. doi: 10.1177/0733464818821787. Epub 2019 Jan 9. PMID 30623709
- [Background] Takizawa C, Gemmell E, Kenworthy J, Speyer R. A Systematic Review of the Prevalence of Oropharyngeal Dysphagia in Stroke, Parkinson's Disease, Alzheimer's Disease, Head Injury, and Pneumonia. Dysphagia. 2016 Jun;31(3):434-41. doi: 10.1007/s00455-016-9695-9. Epub 2016 Mar 12. PMID 26970760